CLINICAL TRIAL: NCT01150188
Title: Effects of Amino Acids on Regional Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 139210; 1R01AG033761-01A1 (NIH)
Record Dates: First submitted 2010-06-22; First posted 2010-06-24 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hypertriglyceridemia
Keywords: aging; lipid metabolism; very low density lipoproteins; amino acids; dietary supplements
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amino acids (Active Comparator): Amino acid supplementation between meals for eight weeks
  Interventions: Dietary Supplement: Amino acids
- Placebo (Placebo Comparator): Supplementation of placebo (inert components) between meals for eight weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Amino acids — 11 g amino acids two times per day for eight weeks
  Arms: Amino acids
Dietary Supplement: Placebo — Placebo of inert compounds, 11 g two times per day for eight weeks
  Arms: Placebo

SUMMARY:
Elevated fat level in blood is a risk factor for coronary heart disease, a major cause of death in America. The overall goal of this project is to test a novel treatment using nutrient (amino acid) supplementation against this condition in men and women, and to understand how this treatment works.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) remains the single largest killer of American men and women (45). Hyper¬triglyceridemia (elevated triglyceride [TG] concentration in the blood) has been shown to be a significant independent risk factor for CHD (7;8;25), accordingly, treatment for hypertriglyceridemia has been included in the Adult Treatment Panel III (ATP III) of the National Cholesterol Education Program (36). In a meta-analysis of 21 population-based prospective studies including a total of 65,863 men and 11,089 women, each increase of 89 mg/dl (1 mmol/l) in TG concentration was associated with a 32% increase in CHD risk in men and 76% increase in women (3). Thus, hypertriglyceridemia is an even stronger risk factor for CHD in women than in men.

The prevalence of hypertriglyceridemia is high. It is a common finding with aging, and is also associated with overweight, obesity, diabetes, and renal disease (39). With the aging of the US population and ongoing epidemics of obesity and type 2-diabetes, the number of individuals with conditions associated with elevated TG levels is likely to grow.

4.1.2 Effect of Amino Acids on Plasma Triglyceride Concentration In an effort to clarify the potential independent effect of protein on plasma and tissue lipids, we supplemented a normal weight-maintaining diet with a relatively small amount of amino acids (~90 kcal/day) between meals. We measured tissue lipids in addition to plasma lipids since the increase in insulin resistance with aging has been linked to increased fat accumulation in muscle and liver tissue (20;63). Also, it has repeatedly been shown that amino acid intake stimulates muscle protein synthesis and improves muscle protein net balance (86). Our hypothesis was that supplementation of the normal diet with a mixture of amino acids will reduce circulating and tissue TG concentrations and improve insulin sensitivity in elderly subjects with impaired glucose tolerance. Twelve impaired glucose tolerant elderly ingested 11 g of essential amino acids (EAA) + arginine twice a day for 16 weeks, after a 7 week control run in. Diet and activity were not otherwise modified. We found individuals consuming the EAA supplement had improved physical function. Further, these individuals had lower plasma and liver TG concentrations than before supplementation, and total cholesterol and VLDL-cholesterol concentrations were also lower after supplementations (12). In the present study, we will investigate this by supplementing the diet of older subjects shown to have hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years.
* Men and Women (Women postmenopausal).
* Ability to sign informed consent, including ≥26 Mini-Mental State Exam.
* Plasma triglyceride concentration between 130-500 mg/dl.

Exclusion Criteria:

* Diabetes (plasma glucose: fasting ≥126 mg/dl or ≥200 mg/dl at 2 hr after 75 g glucose load).
* On diabetes medication or lipid altering agents, including over the counter fish oil/omega 3 fatty acids.
* Kidney/renal or liver disease.
* Bleeding disorders or anemia.
* Endocrine disease.
* Positive hepatitis or HIV screens.
* Alcohol abuse or drug abuse
* Score of <26 on the Mini-Mental State Exam.
* Allergy to iodine or fish products.
* Subjects with cerebral aneurysm clips, internal transistorized devices (e.g., neural stimulators), or cardiac pacemakers.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Very low density lipoprotein (VLDL) turnover | Eight weeks
  Turnover rates of VLDL-triglycerides and VLDL-ApoB-100, including synthesis and breakdown rates, measured before and after eight weeks of amino acid supplementation

SECONDARY OUTCOMES:
Fat oxidation | 8 weeks
  Fat oxidation measured before and after eight weeks of amino acid supplementation
Lipolysis | 8 weeks
  Lipolysis measured before and after eight weeks of amino acid supplementation
Triglyceride uptake in muscle and adipose tissue | Eight weeks
  Triglyceride uptake in muscle and adipose tissue measured before and after eight weeks of amino acid supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Science, Reynolds Aging Institute, Little Rock, Arkansas, United States